# STATISTICAL ANALYSIS PLAN: INDV-2000-102 Part III

**Protocol Title:** A Phase I Double-Blind, Placebo-Controlled Randomized Study to Assess Repeated Doses of INDV-2000 (C4X\_3256) up to 28 Days in Healthy Volunteers, and an Open-Label Study of INDV-2000 up to 11 Days in Treatment Seeking Individuals with Opioid Use Disorder

Final Version: 04 Dec 2023

**NCT:** NCT04976855

# Statistical Analysis Plan

**Protocol Title:** A Phase I Double-Blind, Placebo-Controlled Randomized

Study to Assess Repeated Doses of INDV-2000 (C4X\_3256) up to 28 Days in Healthy Volunteers, and an Open-Label Study of INDV-2000 up to 11 Days in Treatment Seeking Individuals

with Opioid Use Disorder

**Protocol Number:** INDV-2000-102

Compound Number: INDV-2000 (C4X\_3256)

**Sponsor Name:** Indivior

Legal Registered Address: 10710 Midlothian Turnpike, Suite 125

North Chesterfield, VA 23235

USA

**IND Number:** 145881

**Protocol Version:** Amendment 4.0, Version 5.0

**Date:** 08 May 2023

#### Confidentiality Statement

The information contained in this document is privileged and confidential. Do not copy, circulate, or otherwise distribute without written authorization from Indivior Inc.

# **Statistical Analysis Plan Approval**



# **TABLE OF CONTENTS**

| STATISTICAL ANALYSIS PLAN | 1 |
|------------------------------------------------|----|
| TABLE OF CONTENTS | 3 |
| LIST OF TABLES | 5 |
| LIST OF FIGURES | 5 |
| 1. INTRODUCTION | 6 |
| VERSION HISTORY | 6 |
| 1.1. Objectives and Endpoints | 6 |
| 1.2. Study Design. | 10 |
| 2. STATISTICAL HYPOTHESES | 10 |
| 2.1. Multiplicity Adjustment | 11 |
| 3. SAMPLE SIZE DETERMINATION | 11 |
| 4. POPULATIONS FOR ANALYSIS | 11 |
| 5. STATISTICAL ANALYSES | 11 |
| 5.1. General Considerations | 11 |
| 5.1.1. Timing of Analyses | 11 |
| 5.1.2. Programming Environment | 12 |
| 5.1.3. Reporting Conventions | 12 |
| 5.1.4. General Analysis Conventions | 12 |
| 5.1.5. Definitions. | 12 |
| 5.2. Study Conduct and Participant Disposition | 13 |
| 5.3. Primary Endpoints Analysis | 14 |
| 5.3.1. Definition of Endpoints | 14 |
| 5.3.2. Main Analytical Approach | 14 |
| 5.4. Exploratory Endpoints Analysis | 14 |
| 5.4.1. Definition of Endpoints | 14 |
| 5.4.2. Main Analytical Approach | 14 |
| 5.5. Other Safety Analyses | 15 |
| 5.5.1. Extent of Exposure | 15 |
| 5.5.2. Adverse Events | 15 |
| 5.5.3. Additional Safety Assessments | 16 |
| 5.5.3.1. Laboratory Data | 16 |
| 5.5.3.2. Vital Signs | 17 |

| 5.5.3.3. Electrocardiogram (ECG) Data | 18 |
|-------------------------------------------------------------------|----|
| 5.5.3.4. Columbia-Suicide Severity Rating Scale (C-SSRS) | 18 |
| 5.6. Other Analyses | 18 |
| 5.6.1. Demographic and Baseline Characteristics | 18 |
| 5.6.2. Medical History | 19 |
| 5.6.3. Prior and Concomitant Medications and Therapies | 19 |
| 5.6.4. Protocol Deviations | 19 |
| 5.7. Interim Analyses | 19 |
| 6. SUPPORTING DOCUMENTATION | 19 |
| 6.1. Appendix 1: List of Abbreviations | 20 |
| 6.2. Appendix 2: Changes to Protocol-Planned Analyses | 21 |
| 6.3. Appendix 3: Definition and Use of Visit Windows in Reporting | 21 |
| 6.4. Appendix 4: Endpoint Derivations | 21 |
| 6.4.1. Pharmacokinetic Endpoints | 21 |
| 6.4.2. Pharmacodynamic Endpoints. | 21 |
| 6.4.2.1. | 21 |
| 6.4.2.2. | 22 |
| 6.4.2.3. | 22 |
| 6.4.2.4. | 23 |
| 6.4.2.5. | 23 |
| 6.4.3. Safety Endpoints | 23 |
| 6.4.3.1. | 23 |
| 6.5. Appendix 5: Statistical Methodology Details | 23 |
| 6.5.1. PK Analysis | 23 |
| 6.5.1.1. Concentration | 23 |
| 6.5.1.2. PK Parameters | 24 |
| 6.6. Appendix 6: Methods to Manage Missing Data | 24 |
| 6.6.1. Rule for Missing Pre-dose Concentrations | 24 |
| 6.6.2. Missing Pre-dose Sampling Date/Times | 25 |
| 6.6.3. BLQ Concentrations | 25 |
| 6.6.4. Exposure | 25 |
| 6.6.5. AEs | 25 |
| 6.6.6. Medications and Therapies | 26 |

| 6.7. Appendix | x 7: Data Set Descriptions | 27 |
|---------------|--------------------------------|----|
| 7. REFEREN | ICES | 27 |
| | LIST OF TABLES | |
| Table 1 | SAP Version History Summary | 6 |
| Table 2 | Study Objectives and Estimands | 7 |
| Table 3 | Analysis Populations | 11 |
| Table 5 | Planned Laboratory Evaluations | 17 |
| | LIST OF FIGURES | |
| Figure 1. | Study Schematic | 10 |

#### 1. INTRODUCTION

This statistical analysis plan (SAP) provides the detailed methodology for summary and statistical analyses of the data collected in Study INDV-2000-102 Part III and is based on Protocol Amendment 4/09 May 2023 (Version 5.0). This SAP supersedes the statistical considerations stated in the protocol; any differences are identified in <u>Appendix 2</u> of this document. However, major modifications of the primary endpoint definition or its analysis will also be reflected in a protocol amendment. Post hoc or unplanned analyses not specified in the SAP will be documented in the clinical study report (CSR).

#### VERSION HISTORY

Table 1 SAP Version History Summary

| SAP<br>Version | SAP<br>Finalization<br>Date | Associated<br>Protocol<br>Amendment | Protocol<br>Approval<br>Date | Change | Rationale |
|---|---|---|---|---|---|
| 1.0 | 04Dec2023 | Amendment<br>4.0,<br>Version 5.0 | 09May2023 | Not Applicable | Original version |

#### 1.1. Objectives and Endpoints

Each study objective is presented in <u>Table 2</u> with associated estimands. Intercurrent events occur after treatment starts and either preclude the observation of an endpoint or affect its interpretation. For the intercurrent event of study discontinuation, the principal stratum strategy will be used for pharmacokinetic (PK) endpoints in that only subjects with an adequate amount of PK data will be included in the PK population; for all other endpoints, the while-on-treatment strategy will be used since data will be collected only up to end of study (EOS) or study discontinuation. Other potential intercurrent events in this study are prohibited medications and lifestyle restrictions detailed in protocol sections 9.6.2 and 9.6.3, respectively. Possible strategies for these intercurrent events are treatment policy (intercurrent event is ignored), while on treatment (data collected after the event is ignored), and principal stratum for PK endpoints (subject is excluded from the PK population), to be decided by the sponsor on a case-by-case basis.

 Table 2
 Study Objectives and Estimands

| | | Estimand | • | |
|---|---|---|---|---|
| Objective<br>Clinical Category | Statistical<br>Category | Variable/Endpoint | Pop-<br>ulation | Population-Level Summary |
| Primary Objective Assess the safety and to opioid use disorder (OU | • | ng repeated doses of INDV-2000 administered alone and with String population. | UBOXON | E sublingual (SL) film in an |
| Adverse Events (AEs) | Primary | Incidence, severity, and relatedness of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs) and events leading to study discontinuation or death. | Safety | Categorical descriptive |

Exploratory Objectives

| | | Estimand | | |
|---|---|---|---|---|
| Objective<br>Clinical Category | Statistical<br>Category | Variable/Endpoint | Pop-<br>ulation | Population-Level Summary |

| | | Estimand | | |
|---|---|---|---|---|
| Objective<br>Clinical Category | Statistical<br>Category | Variable/Endpoint | Pop-<br>ulation | Population-Level Summary |
| omneur outegory | | 1 | | |

#### 1.2. Study Design

This is a Phase I study to assess repeated doses of INDV-2000 in healthy volunteers and in treatment-seeking individuals with OUD. The study will be conducted in three parts, as depicted in <u>Figure 1</u>. This SAP is for Part III only.

Figure 1. Study Schematic



Key features of the study design are described below.

- Part III is an open-label study in OUD treatment-seeking individuals.
- Part III dose determination will follow a blinded review of safety and PK data from Parts I and II.
- The screening period for Part III is up to 35 days. Subjects will receive SUBOXONE SL film during a 6-day, in-clinic run-in period. Qualifying subjects will then be enrolled into the study, consisting of a 14-day in-clinic period followed by an EOS visit on Day 21. Subjects will receive SUBOXONE SL film alone on Days 1 and 2, SUBOXONE SL film and INDV-2000 on Days 3-9, and INDV-2000 alone on Days 10-13. Total study duration per subject, from screening through the EOS visit, will be approximately 56 days.

#### 2. STATISTICAL HYPOTHESES

There will be no statistical inference in this study. All statistics will be descriptive only.

#### 2.1. Multiplicity Adjustment

There will be no statistical inference in this study; therefore, there will be no need for multiplicity adjustment.

#### 3. SAMPLE SIZE DETERMINATION

The sample size for each part of the study is not based on formal power calculations because the study is designed to provide preliminary descriptive assessments of the safety, tolerability and PK for INDV-2000. The sample sizes used are typical for studies of this nature and should be adequate to assess the parameters described.

#### 4. POPULATIONS FOR ANALYSIS

Data for all subjects will be assessed to determine if subjects meet the criteria for inclusion in each analysis population shown in <u>Table 3</u> prior to releasing the database and classifications will be documented per standard operating procedures.

**Table 3** Analysis Populations

| Population | Description |
|---|---|
| Screened | Subjects who signed informed consent. |
| Enrolled | Subjects who met Day -1 run-in assessment criteria. |
| Safety | Subjects who received at least one dose of investigational |
| | medicinal product (IMP). Subjects will be summarized |
| | according to the study treatment received. |
| Run-In Safety | Subjects who received at least one dose of study drug during the run-in period. |
| PK | Subjects who received at least one dose of INDV-2000, have an adequate number of PK samples collected to derive any PK parameter, and have no protocol deviations that would significantly alter plasma concentration of INDV-2000. |

#### 5. STATISTICAL ANALYSES

#### 5.1. General Considerations

# **5.1.1.** Timing of Analyses

Database lock and final production of tables, figures, and listings (TFLs) will occur after the completion of Part III.

#### 5.1.2. Programming Environment

SAS® version 9.4 or higher (SAS Institute, Cary, North Carolina) will be used for statistical analyses and for the production of Study Data Tabulation Model (SDTM) and Analysis Data Model (ADaM) data sets as well as TFLs.

#### 5.1.3. Reporting Conventions

Data will be summarized by visit for visit-based assessments and by treatment for non-visit-based assessments, if applicable. TFL tables of contents, mock-ups, and specifications are provided in a separate document from the SAP. The following reporting conventions will be followed:

- Treatment group names and order in tables and figures for non-visit-based assessments, where applicable, will be SUBOXONE, INDV-2000+SUBOXONE, INDV-2000, All Subjects; some of these tables may omit the All Subjects groups. Tables and figures for visit-based assessments will only show All Subjects and will include a footnote to describe treatments administered for each visit, if applicable.
- Tables and figures will present summaries/analyses by study visit and time point, if applicable, for visit-based assessments.
- Table column headers and figure legends will include subgroup sample sizes ("N = xx"). Sample sizes reported as part of descriptive statistics ("n") will be the number of non-missing observations.
- Listings will generally include unique subject identifier (including site identifier); treatment, if applicable, if the assessment is not visit-based; study visit/time point; assessment or collection date/time; parameter; and observed value.

#### 5.1.4. General Analysis Conventions

Categorical variables will be summarized using frequencies and percentages. Percentages will be reported to one decimal place.

Continuous variables will be summarized using descriptive statistics (e.g., n, mean, standard deviation (SD), distribution percentiles, range). The number of decimal places for minimums and maximums will be the same as the source data. The number of decimal places for means, medians, and interquartile ranges will be the same as the source data plus one, and the number of decimal places for measures of variance will be the same as the source data plus two. See Section 6.5 (Appendix 5) for summary statistics and precision specifications for PK data.

Data with qualifiers (e.g., "<") will be listed with but summarized without the qualifier.

#### **5.1.5. Definitions**

IMP: INDV-2000 or placebo (placebo not applicable in Part III)

Study Drug: INDV-2000, SUBOXONE SL film, or placebo (placebo not applicable in Part III).

<u>Screening Period</u>: Informed consent to Day -7 Clinic Check-In.

Run-In Period: Day -7 to Day -1 Run-In Assessment

End-of-Study (EOS): Early termination or completion of last scheduled visit.

Enrolled Subject: Met Day -1 run-in assessment criteria.

Study Day 1: day of first dose of study drug administration after the run-in period.

#### Study day:

- Study day = date of assessment date of Study Day 1 + 1, for assessments on or after Study Day 1
- Study day = date of assessment date of Study Day 1, for assessments before Study Day 1

Study time: time of assessment – time of first study drug administered in the clinical unit.

#### Duration:

- Duration in days = end date start date + 1
- Duration in minutes = end time start time. Durations will be adjusted for Daylight Saving Time, where applicable.

<u>Baseline observation</u>: for a given parameter for a given subject, the last observed value, including unscheduled and repeated assessments, before the first dose of IMP or planned first dose of IMP if IMP was not administered.

<u>Run-in baseline observation</u>: for a given parameter for a given subject, the last observed value, including unscheduled and repeated assessments, before the first dose of study drug during the run-in period.

#### 5.2. Study Conduct and Participant Disposition

Subject disposition summaries will include the number of subjects who were screened for Part III, who were screen failures, who were run-in failures, who were enrolled, who were in each analysis population, and who completed the study. For percentages, the number of subjects screened will be the denominator for screen and run-in failures and for the Run-In Safety Population, which in turn will be the denominator for subjects enrolled. The number of subjects enrolled will be the denominator for the Safety and PK analysis populations and for subjects completing the study.

Reason for study discontinuation will be summarized by number and percentage of subjects for each reason reported; for the percentage, the number of subjects who discontinued will be the denominator.

Reason for screen failure will be summarized in a separate table by number and percentage of subjects for each reason reported; the denominator will be the number of screen failures.

#### 5.3. Primary Endpoints Analysis

#### 5.3.1. Definition of Endpoints

The primary endpoints are incidence of TEAEs, maximum severity TEAEs, TEAEs related to study drug, treatment-emergent serious adverse events (TESAEs), and TEAEs leading to study discontinuation or death.

#### 5.3.2. Main Analytical Approach

Estimand strategy: While on treatment.

Analysis set: Safety (see Table 3).

Analysis methodology: Descriptive only.

Intercurrent events and missing data: AE data will no longer be collected on subjects who discontinue early from the study except as required to resolve an ongoing AE. See <u>Section 6.6.3 (Appendix 6)</u> for details on handling of missing AE information.

See Section 5.6.2 for details on AE summaries and listings.

#### 5.4. Exploratory Endpoints Analysis

# 5.4.1. Definition of Endpoints

#### 5.4.2. Main Analytical Approach





#### 5.5. Other Safety Analyses

#### 5.5.1. Extent of Exposure

Study drug exposure will be summarized as total number of doses and dose duration (days), separately for INDV-2000 (Safety Population) and buprenorphine (Run-In Safety Population). For INDV-2000, exposure will be summarized for study days 3-9 (with buprenorphine), study days 10-13 (without buprenorphine) and study days 3-13. For buprenorphine, exposure will be summarized for run-in, study days 1-2 (without INDV-2000), study days 3-9 (with INDV-2000), and study days 1-9.

#### 5.5.2. Adverse Events

A TEAE is an AE that started at or after first administration of IMP. A run-in AE is an AE that started at or after first administration of study drug during the run-in period. AEs will be assigned to study treatments based on start dates and times of treatments and start dates and times of AEs.

AEs will be coded to a System Organ Class (SOC) and Preferred Term (PT) using Medical Dictionary for Regulatory Activities (MedDRA). Additional details of the coding process, including the current version of the dictionary, are described in the Data Management Plan. All AEs will be listed for individual subjects. Listings will include SOC, PT, and reported term; treatment; onset date and time, end date, and duration; run-in status, treatment-emergence, severity, toxicity grade (though not required for Part III of the study), seriousness and seriousness criteria; relationship to study drug; action taken with IMP; action taken with SUBOXONE SL film; whether concomitant treatment was given; outcome; and whether the AE resulted in study discontinuation. Duration (days) is calculated as the AE end date – the AE onset date +1; for ongoing AEs, the date of end of study participation will be used as the end date. Duration will be missing if either the start or end date is partially or completely missing. SAEs, TEAEs leading to IMP discontinuation or interruption, AEs leading to SUBOXONE SL film discontinuation or interruption, and fatal AEs will be listed separately.

The incidence and number of all TEAEs, TESAEs, study drug-related TEAEs and TESAEs, severe TEAEs, TEAEs leading to IMP discontinuation or interruption, and fatal TEAEs will be presented in an overall summary table.

TEAEs, TESAEs, study drug-related TEAEs and TESAEs, and run-in AEs will be summarized by MedDRA SOC and PT, each in descending order of frequency among all subjects within study part (then alphabetically in case of ties). TEAEs will also be

summarized by maximum severity within SOC and PT. If an AE is reported more than once by a subject within a SOC and/or PT, the maximum reported level of severity will be used at each level of summation in the severity summary table.

Incidence and number of TEAEs will also be summarized by PT only (ie, not SOC), sorted by descending frequency among all subjects (within study part).

Non-treatment-emergent, non-run-in AEs are defined as AEs that started either before first administration of study drug or after the run-in period but before first administration of IMP and will be summarized for the run-in safety population.

See Section <u>6.6.3</u> (Appendix 6) for details on handling of missing AE information.

#### 5.5.3. Additional Safety Assessments

#### 5.5.3.1. Laboratory Data

Planned laboratory evaluations (<u>Table 5</u>) will be summarized by analysis visit as observed values and, for numeric values, changes from baseline. Normal/abnormal shifts from baseline will also be summarized. Abnormal laboratory evaluations will be listed separately. Laboratory evaluations done only at screening and during run-in will be listed but not summarized, unless included as baseline observation. Reported values of clinical laboratory parameters that include qualifiers (ie, <,  $\le$ , >,  $\ge$ ) will be listed as reported but will be summarized without the qualifier.

#### **Table 4** Planned Laboratory Evaluations

Haematology
Haematocrit
Serum Chemistry:
Albumin

Haemoglobin Alkaline phosphatase

Mean corpuscular haemoglobin Alanine aminotransferase (ALT)

Mean corpuscular haemoglobin concentration Amylase

Mean corpuscular volume Aspartate aminotransferase (AST)

Platelet count Blood urea nitrogen

Red blood cell count
White blood cell count with differential (absolute count)
Carbon dioxide

White blood cell count with differential (absolute count)

Carbon dioxide
Chloride

Urinalysis:

Creatinine

Appearance Creatine kinase
Bilirubin Gamma-glutamyl transferase
Colour Glucose (non-fasting)

Glucose Lactate dehydrogenase Lipase

Leucocyte esteraseMagnesiumMicroscopic examination of sedimentaPhosphorusNitritePotassiumOccult bloodSodiumpHTotal bilirubin

Protein Direct bilirubin
Specific gravity Total cholesterol
Urobilinogen Total protein

Triglycerides

Pregnancy:

Serum hCG Urine Drug Screen (UDS):

Urine hCG Opioids
Cocaine
Molecular Amphetamines

PCR for COVID-19

Cannabinoids
Barbiturates
Screening Only:

Benzodiazepines

FSH (as needed in post-menopausal females only)

Haemoglobin A1c

Hepatitis B surface Antigen

Methamphetamine
Phencyclidine
Ethanol

Hepatitis C Antibody In addition to the above, for Part III:

HIV-1 and -2 antibodies Fentanyl
Prothombin Time with INR Oxycodone

PTT

Anti-HIV = human immunodeficiency virus antibodies; hCG = human chorionic gonadotropin; INR = international normalized ratio; and PTT = partial thromboplastin time.

#### **5.5.3.2. Vital Signs**

Vital signs (systolic and diastolic blood pressure, heart rate, respiratory rate, temperature) will be summarized as observed values and changes from baseline by analysis visit and time point. Vital signs during the run-in period will be summarized separately.

<sup>&</sup>lt;sup>a</sup> Microscopic examination of sediment will be performed only if the results of the urinalysis evaluation are positive (microscopic examination may include but is not limited to White Blood Cell count, Red Blood Cell count, casts and crystals).

#### 5.5.3.3. Electrocardiogram (ECG) Data

Numeric 12-lead ECG parameters [heart rate, PR interval, QRS duration, QT interval, Fridericia's corrected QT interval (QTcF)] will be summarized as observed values and changes from baseline by analysis visit and time point. ECG interpretation (normal, abnormal not clinically significant, abnormal clinically significant) will be summarized by visit and time point as shifts from baseline.

#### **5.5.3.4.** Columbia-Suicide Severity Rating Scale (C-SSRS)

The composite endpoints Suicidal Ideation and Suicidal Behavior will be derived from the following 10 binary C-SSRS questions, reordered from the actual scale to facilitate the derivation:

| Question 1 | Wish to be Dead |
|---|---|
| Question 2 | Non-specific Active Suicidal Thoughts |
| Question 3 | Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act |
| Question 4 | Active Suicidal Ideation with Some Intent to Act, without Specific Plan |
| Question 5 | Active Suicidal Ideation with Specific Plan and Intent |
| Question 6 | Preparatory Acts or Behavior |
| Question 7 | Aborted Attempt |
| Question 8 | Interrupted Attempt |
| Question 9 | Actual Attempt (non-fatal) |
| Question 10 | Completed Suicide |

Suicidal Ideation is derived as "yes" if any of Question 1-5 has a "yes" response. Suicidal Behavior is derived as "yes" if any of Question 6-10 has a "yes" response. If there are zero "yes" responses and at least one question has a missing response, the derived composite will be missing. Suicidal Ideation and Suicidal Behavior will be summarized as categorical variables by analysis visit.

#### 5.6. Other Analyses

#### 5.6.1. Demographic and Baseline Characteristics

Demographic and other baseline characteristics will be summarized separately for the run-in safety, safety, and PK populations, if different. Parameters to be summarized will be age, sex, race, ethnicity, fertility status, height/weight/body mass index, and substance use (alcohol, nicotine, xanthine/caffeine) status (never/current/former). Listings will include all subjects, including screen failures and run-in failures.

#### 5.6.2. Medical History

Relevant medical history will be coded using MedDRA (refer to the Data Management Plan) and will be listed for the run-in safety population.

#### 5.6.3. Prior and Concomitant Medications and Therapies

Medications and therapies will be collected from screening through EOS and will be coded using Anatomical Therapeutic Chemical (ATC) classification codes via the World Health Organization Drug Dictionary (WHO-DD). Additional details of the coding process, including the current version of the dictionary, are described in the Data Management Plan. Prior medications and therapies will be medications/therapies that ended before first administration of study drug or were taken by subjects who did not take study drug. Therapies and medications that were started or were ongoing during run-in will be considered run-in therapies and medications. Therapies and medications that were started or were ongoing post run-in will be considered concomitant therapies and medications. A therapy or medication can be both run-in and concomitant. Therapies/medications will be assigned to study treatments based on start dates and times of treatments and start and end dates and times of therapies/medications.

Prior concomitant medications and therapies will be summarized for all subjects. Run-in medications and therapies will be summarized for the run-in safety population. Concomitant medications and therapies will be summarized for the safety population. The summary of incidence (number and percentage of subjects reporting the medication/therapy at least once) will be sorted alphabetically by therapeutic class (ATC level 2) and standardized medication/therapy name.

See Section <u>6.6.4 (Appendix 6)</u> for details on handling missing information on medications and therapies.

#### 5.6.4. Protocol Deviations

Protocol deviations will be identified and documented prior to database lock and will be summarized by category (eg, prohibited medication, out-of-window assessment) and type (eg, major, minor), per the Protocol Deviation Plan for the study, for the run-in safety population. Deviations that occur in subjects who were not dosed with study drug, if any, will be summarized separately. All protocol deviations will be listed.

#### 5.7. Interim Analyses

Not applicable.

#### 6. SUPPORTING DOCUMENTATION

# 6.1. Appendix 1: List of Abbreviations

| Abbreviation | Term |
|--------------|----------------------------------------------|
| ADaM | Analysis Data Model |
| AE | adverse event |
| ATC | Anatomic Therapeutic Chemical |
| BLQ | below limit of quantitation |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| CRF | Case Report Form |
| CSR | clinical study report |
| ECG | electrocardiogram |
| EOS | end of study |
| h | hours |
| IMP | investigational medicinal product |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mm | millimeter |
| OUD | opioid use disorder |
| PK | pharmacokinetic |
| PT | Preferred Term |
| QTcF | Fridericia's corrected QT interval |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SD | standard deviation |
| SDTM | Study Data Tabulation Model |
| SL | sublingual |
| SOC | System Organ Class |
| TEAE | |
| TEAE | treatment-emergent adverse event |
| TESAE | treatment-emergent serious adverse event |
| TFLs | tables, figures, and listings |
| WHO DD | World Hoolth Organization Deva Dictionary |
| WHO-DD | World Health Organization Drug Dictionary |

# 6.2. Appendix 2: Changes to Protocol-Planned Analyses

The following are changes from the protocol that are in the SAP:

| Protocol: | SAP: |
|-----------|-------------------------------------|
| | Added Screened analysis population. |
| | Added Enrolled analysis population. |

# 6.3. Appendix 3: Definition and Use of Visit Windows in Reporting

No windowing will be used for summaries. Analysis visits will be visits denoted in the Case Report Form (CRF). If a subject has more than 1 assessment for a given visit, the most recent non-missing assessment will be used for summaries.

# 6.4. Appendix 4: Endpoint Derivations

6.4.1. Pharmacokinetic Endpoints

#### 6.4.2. Pharmacodynamic Endpoints







# 6.4.3. Safety Endpoints

# 6.5. Appendix 5: Statistical Methodology Details

Statistical programming will be done using SAS version 9.4 (or later) on a Windows 10 Enterprise (or later) operating system. Plasma PK parameters will be calculated using Phoenix<sup>TM</sup> WinNonlin<sup>®</sup> (Version 8.3.4, Certara, LP).

# 6.5.1. PK Analysis

# 6.5.1.1. Concentration



| 6.5.1.2. PK Parameters |
|-------------------------------------------------|
| 6.6. Appendix 6: Methods to Manage Missing Data |
| 6.6.1. Rule for Missing Pre-dose Concentrations |

#### 6.6.2. Missing Pre-dose Sampling Date/Times

If a missing pre-dose concentration is also missing sampling date/time (due to the sample not being drawn), the sampling date/time will be imputed with the corresponding dosing date/time on that day.

#### 6.6.3. BLQ Concentrations

Concentration values that are reported as BLQ will be presented as "BLQ" in concentration listings, replaced by 0 for summary statistic calculations and linear-scale plots of concentrations, and excluded from semi-logarithmic-scale plots of concentrations.

For derivations of PK plasma parameters, all concentrations that are BLQ prior to the first measurable concentration will be set to zero. BLQ values that are between measurable concentrations will be set to missing. Measurable concentrations immediately between 2 BLQ values will be set to missing. Measurable concentrations following two or more consecutive BLQ concentrations will be set to missing. The BLQ values following the last quantifiable time points will be set to missing. No concentration estimates will be imputed for missing sample values.

#### 6.6.4. Exposure

#### **Missing Study Drug Dosing Information**

All efforts should be made to obtain missing study drug dosing information from the investigator. If data are still missing after all efforts, then total exposure will be missing.

#### Missing Last Date of Study Drug Exposure

All efforts should be made to obtain missing last date of study drug exposure from the investigator. If the last date of exposure is still missing after all efforts, then the last available dosing record date may be used as the last study drug exposure date for the calculation of exposure duration.

#### 6.6.5. AEs

#### **Missing AE Severity**

Missing AE severity must be queried until resolution. In the unlikely event that resolution is not possible, missing severity will be imputed as "severe" in summaries.

## Missing AE Relationship to Study Drug

Missing relationship to study drug for a TEAE must be queried until resolution. In the unlikely event that resolution is not possible, missing relationship will be imputed as "related" in summaries.

#### **Missing AE Seriousness**

Missing AE seriousness must be queried until resolution. Seriousness cannot be imputed as "serious" since doing so would affect the reconciliation between the trial database and the SAE registry.

#### Missing AE Start Date/Time Information

Note: partial times will not be recorded in the CRF.

An AE will be considered a run-in AE for the Run-In Safety Population under the following conditions:

- Missing start year, month, day, time and it can be deduced from non-missing components of AE end date that the AE ended before first IMP.
- Missing start month, day, time if start year is equal to or after year of first study drug during run-in and it can be deduced from non-missing components of AE end date that AE ended before first IMP.
- Missing start day and time if start year is after year of first study drug during run-in or if start year is equal to year of first study drug during run-in and month is equal to or after month of first study drug during run-in and it can be deduced from non-missing components of AE end date that AE ended before first IMP.
- Missing start time if start date is on or after date of first study drug during run-in and it
  can be deduced from non-missing components of AE end date that AE ended before first
  IMP.

An AE will be considered treatment emergent for the Safety Population under the following conditions:

- Missing start year, month, day, time unless it can be deduced from non-missing components of AE end date that the AE ended before first IMP.
- Missing start month, day, time if start year is equal to or after year of first IMP, unless it can be deduced from non-missing components of AE end date that AE ended before first IMP.
- Missing start day and time if start year is after year of first IMP or if start year is equal to year of first IMP and month is equal to or after month of first IMP, unless it can be deduced from non-missing components of AE end date that AE ended before first IMP.
- Missing start time if start date is on or after date of first IMP.

#### **6.6.6.** Medications and Therapies

#### Missing End Date/Time Information

Note: partial times will not be recorded in the CRF.

Run-in and concomitant status will be assigned as follows:

A medication/therapy will be considered run-in under the following conditions:

- Missing end year, month, day, time and it can be deduced from non-missing components of the start date that the medication/therapy started before or during run-in.
- Missing end month, day, time if end year is equal to or after start year of run-in and it can be deduced from non-missing components of the start date that the medication/therapy started before or during run-in.
- Missing end day and time if end year/month is equal to or after start year/month of run-in and it can be deduced from non-missing components of the start date that the medication/therapy started before or during run-in.
- Missing end time if end date is on or after start date of run-in and it can be deduced from non-missing components of the start time that the medicaton/therapy started before or during run-in.

A medication/therapy will be considered concomitant under the following conditions:

- Missing end year, month, day, time and it can be deduced from non-missing components of the start date that the medication/therapy started before or during post run-in.
- Missing end month, day, time if end year is equal to or after start year of post run-in and it can be deduced from non-missing components of the start date that the medication/therapy started before or during post run-in.
- Missing end day and time if end year/month is equal to or after start year/month of post run-in and it can be deduced from non-missing components of the start date that the medication/therapy started before or during post run-in.
- Missing end time if end date is on or after start date of post run-in and it can be deduced from non-missing components of the start time that the medicaton/therapy started before or during post run-in.

#### 6.7. Appendix 7: Data Set Descriptions

Trial data sets will consist of CRF exports and external data files. External files may be used for protocol deviations and data from the central laboratory, for example.

## 7. REFERENCES

None.